CLINICAL TRIAL: NCT01077687
Title: Expanding Rapid Ascertainment Networks of Schizophrenia Families in Taiwan
Acronym: S-TOGET
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Collaborators: University of California, San Diego (Other)
Responsible Party: Sponsor
Other Study IDs: 200810016R; U.S. NIH Grant1R01MH085560-01 (Other Grant/Funding Number: U.S. NIH Grant/Contract Award Number)
Record Dates: First submitted 2010-02-25; First posted 2010-03-01 (Estimated); Last update posted 2021-02-08 (Actual); Status verified 2021-02

CONDITIONS: Schizophrenia
Keywords: schizophrenia; genome-wide association study (GWAS); single-nucleotide polymorphisms (SNPs); Han Chinese population; trio families; Schizophrenia with trio families
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood.
Oversight: Data Monitoring Committee: No

SUMMARY:
This proposal responds to Request for Applications RFA ( Rapid Founding Award)-MH ( Mental Health)-08-131, which seeks applications that propose to enrich pre-existing resources for schizophrenia in the NIMH ( National Institute of Mental Health) Human Genetics Initiative and to apply genomic methods to further our understanding of the molecular etiology of the disorder. The overarching aims of this proposal are to quickly and cost-effectively ascertain a large sample of trio families affected by schizophrenia, and to discover causal variants for the disorder in the first family-based genome-wide association study (GWAS) of the disorder. In Taiwan, there is no such kind of policy to support this kind of GWAS study as it is a very expensive study, including collecting large family samples and genome-wide SNP scanning. We, thus, collaborate with Professor Ming T, Tsuang and his extended subcontracted researchers to apply for this project. We, the research team in Taiwan, will collect 3800 trio families (11400 subjects) of schizophrenia. In our recently completed NIMH-funded Genetic Linkage Study of Schizophrenia (R01MH059624; USA PI: Ming T. Tsuang; Taiwan PI: Hai-Gwo Hwu), the investigators established a large and efficient ascertainment network and infrastructure in Taiwan, which will again be utilized and expanded in the proposed study. Through additional ascertainment within this framework, the investigators will collect an aggregate sample with adequate power for detecting in a GWAS those variants that make even small contributions to the risk for the disorder.

The investigators will meet the overarching goals of this project by accomplishing several Specific Aims, as follows:

1. Rapidly ascertain schizophrenia trio families from ten Taiwanese clinical ascertainment sites;
2. Supplement NIMH Genetics Initiative collections by sending all clinical data and biomaterials to the appropriate repositories;
3. Assess the association of schizophrenia with a genome-wide panel of single-nucleotide polymorphisms (SNPs) and their constituent haplotypes;
4. Analyze quantitative schizophrenia phenotypes such as age at onset ;
5. Perform a genome-wide survey for copy-number variations related to schizophrenia;
6. Test for gene-gene interactions (epistasis); and
7. Test for gene-environment interactions, such as the well-established effect of season of birth.

DETAILED DESCRIPTION:
Over the past four decades, researchers have become increasingly certain that schizophrenia has a complex, multifactorial etiology. Although many twin studies confirm that genes play a substantial role in the etiology of this disabling disorder,5 genome-wide linkage analysis of schizophrenia have produced conflicting results. While many of these studies have identified chromosomal regions showing some evidence for linkage to schizophrenia, no finding has been consistently replicated. Given the high heritability of schizophrenia,5 the failure of linkage methods to find susceptibility genes suggests that these genes each have very small, incremental effects on the expression of the disorder. Risch and Merikangas6 showed that for genes of small effect, the power of linkage studies will be low but the power of association studies will be high. Although meta-analysis of candidate gene association studies have implicated some genes, these findings (even if confirmed by larger studies) would only account for a small fraction of schizophrenia's heritability. These considerations suggest that a genome-wide association scan would be an effective method for finding schizophrenia susceptibility genes. To that end, the investigators have designed a multi-stage analytic plan which involves rapid continued ascertainment of probands and family members from an established clinical ascertainment network in Taiwan, performing a genome-wide association scan (GWAS) on this large sample of affected nuclear families, and pooling the novel GWAS results from this project with those from existing case-control GWAS studies of schizophrenia. To accomplish these objectives, the investigators propose a series of specific aims, as follows:

1. Supplement our previously collected sample of 1,200 Han Chinese schizophrenia-affected nuclear families from Taiwan by rapidly screening and collecting an additional 3,800 trios from eleven ascertainment sites in Taiwan;
2. Assess the association of schizophrenia with a genome-wide panel of single-nucleotide polymorphisms (SNPs) and their constituent haplotypes;
3. Perform a genome-wide survey for copy-number variations related to schizophrenia;
4. Test for gene-gene interactions and epistasis;
5. Test for gene-environment interactions, such as the well-established effect of season of birth;
6. Analyze quantitative schizophrenia phenotypes, such as age at onset; and
7. Enhance the NIMH Genetics Initiative collections by sending all clinical data, biomaterials, and genotypes to the appropriate repositories, and completing a meta-analysis of our family-based GWAS data and those from existing case-control GWASs of schizophrenia in the repository;

The above aims achieve the goals of the RFA in several ways. First, the proposed work would markedly enrich the existing resources of the NIMH Human Genetics Initiative, especially the current pool of schizophrenia-affected nuclear families. Not only would the data and biomaterials from this project enrich the NIMH repositories, the study has been designed to be readily combinable with those already in the repositories to boost the power available for detecting genes with small effects on risk. Further, the proposed project would apply the latest genomic research methods to further our understanding of the molecular etiology of the disorder. Lastly, by capitalizing on an existing clinical infrastructure and an efficient screening and assessment protocol, the investigators will obtain a well-powered sample in a very rapid and cost-effective manner.

ELIGIBILITY:
Inclusion Criteria:

* Schizophrenia
* Trio families (a proband's parents should be recruited)

Exclusion Criteria:

* One or both parents of a proband was not alive
* with mental retardation
* with epilepsy
* with alcohol or substance abuse
* with other organic brain syndromes

Ages: 16 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: schizophrenia Han Chinese Population one sibling with his/her parents
Sampling Method: Non-Probability Sample
Enrollment: 1050 (Actual)
Dates: Start 2009-07; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hai-Gwo Hwu, Professor, Principal Investigator — College of Medicine, National Taiwan University
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan